CLINICAL TRIAL: NCT03585972
Title: Occupational Therapy Services to Improve Frailty Status
Brief Title: Frailty Prevention Program to Prevent Frailty Among Older African Americans
Acronym: FPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Michigan Health Endowment Fund (Other)
Responsible Party: Principal Investigator, Heather Fritz, Assistant Professor of Occupational Therapy and Gerontology, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1701000204
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Frail Elderly Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors do not know which arm participants were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frailty Prevention Program (Experimental): 4 face-to-face sessions, with a licensed and registered occupational therapist over 4 months
  Interventions: Behavioral: Frailty Prevention Program
- Educational materials (No Intervention): Participants receive publicly available educational materials

INTERVENTIONS:
Behavioral: Frailty Prevention Program — 4 face-to-face sessions, with a occupational therapist over 4 months to address function, safety, social participation, diet, exercise, sleep, and medication management. Sessions are expected to last between 60-120 minutes. The first session is a comprehensive occupational therapy evaluation and treatment plan. Sessions 2 and 3 involved physical activity and dietary education, counseling and goal setting. Session 4 involves reviewing program progress, and setting maintenance goals.
  Arms: Frailty Prevention Program

SUMMARY:
Between 20-60% of older adults experience frailty as they age. Frailty is a clinical state of increased vulnerability resulting from aging-associated declines in biological reserve across multiple physiologic systems. Because of the lack of biological reserve, relatively minor physical or psychological assaults have the potential to trigger a cascade of negative sequelae for frail older adults resulting in adverse health outcomes including mortality, disability in basic and instrumental activities of daily living, hospitalization and emergency visits, and institutionalization in community-dwelling older adults. Despite the potential personal and economic consequences of frailty syndrome, frailty is not an irreversible process. For example, a 4.5-year longitudinal study conducted by Gill et al., (2006) demonstrated that of their 754 community dwelling older adults, 58% had at least one change in frailty status during the study period and that approximately one third of these transitions were from a state of greater frailty to one of lesser frailty, suggesting that it is possible to reverse the frailty trajectory. Nonetheless, there is a lack effective means of reversing frailty or slowing the progression of older adults along the frailty continuum.The purpose of the proposed research is to evaluate the feasibility and preliminary effectiveness of an occupational therapy intervention delivered through the primary care setting for improving frailty status and physical functioning among older adults ages 55 and older who are pre-frail when compared to usual care.

DETAILED DESCRIPTION:
Between 20-60% of older adults experience frailty as they age. Frailty is a clinical state of increased vulnerability resulting from aging-associated declines in biological reserve across multiple physiologic systems. Because of the lack of biological reserve, relatively minor physical or psychological assaults have the potential to trigger a cascade of negative sequelae for frail older adults resulting in adverse health outcomes including mortality, disability in basic and instrumental activities of daily living, mobility impairment, falls, hospitalization and emergency visits, and institutionalization in community-dwelling older adults. In addition, frailty results in increased healthcare cost and service utilization across both acute and community settings. Frail older adults (OA) have a higher frequency of primary care visits, consume 50% of all hospital care, use over 80% of home care services, and occupying 90% of all nursing home beds in the United States.

Despite the potential personal and economic consequences of frailty syndrome, frailty is not an irreversible process. For example, a 4.5-year longitudinal study conducted by Gill et al., (2006) demonstrated that of their 754 community dwelling older adults, 58% had at least one change in frailty status during the study period and that approximately one third of these transitions were from a state of greater frailty to one of lesser frailty, suggesting that it is possible to reverse the frailty trajectory. Nonetheless, there is a continued lack effective means of reversing frailty or slowing the progression of older adults along the frailty continuum. Interventions have been developed to slow or reverse frailty and have typically focused on exercise training, nutritional supplementation, pharmaceutical agents, or some combination of those elements. The efficacy of such interventions has been mixed with intensive physical activity interventions demonstrating the most promise. Yet intensive physical activity interventions are difficult to disseminate at a population level, and evidence suggests that even when participants experience a change in their frailty status as a result of intensive exercise intervention, they generally return to their pre-intervention state once exercise training is discontinued. Because of the lack knowledge about how best to address the problem of frailty in older adulthood, researchers have argued that the continued development and evaluation of interventions designed to prevent frailty or ameliorate the consequences of frailty should remain a top priority in aging research.

One approach that holds promise for preventing or slowing the progression of frailty is early identification of pre-frail individuals in the outpatient setting and referring them to occupational therapy services before individuals require more intensive inpatient services. Primary care geriatric clinics afford a unique opportunity for early identification and referral of at risk older adults during the course of routine care. Providers are often times more familiar with their patients, have had the opportunity to track their patient's progress over time, and therefore, are uniquely situated to identify changes in functional or health status and make appropriate referrals on behalf of their patients. While occupational therapists have not traditionally provided services in the primary care setting, occupational therapy services delivered in hospital, home, and community settings improve function and reduce healthcare costs among older adults. Occupational therapy services delivered in the primary care setting offers a unique opportunity to improve the health, function and wellbeing of frail, pre-frail, and at risk older adults (OA).

The purpose of the proposed research is to evaluate the feasibility and preliminary effectiveness of an occupational therapy intervention delivered through the primary care setting for improving frailty status and physical functioning among older adults (OA) ages 55 and older who are pre-frail when compared to usual care. Secondary aims include conducting exploratory analyses to examine potential mechanisms that may explain the intervention's effects, and evaluating the intervention's impact on secondary outcomes including occupational performance, quality of life, and care utilization.

The investigators hypothesize that occupational therapy services will result in greater improvement in the primary outcomes of frailty status (measured via the Fried Frailty criteria), physical function, and the secondary outcomes of occupational performance, health status (measured via weight and blood pressure), and care utilization (assessed via structured questionnaire) Quality of Life among the treatment group compared to usual care. The two specific aims of the study are:

1. To evaluate intervention feasibility and acceptability. Determine if the occupational therapy services delivered are feasible and acceptable. By tracking time, effort, costs, adherence to recommendations, participant recruitment and retention rates, and intervention satisfaction among a sample of 150 pre-frail older adults, we expect to be able to provide data that both support the feasibility of the intervention and help us improve it for a subsequent study.
2. To conduct a pilot randomized trial of the intervention components with 150 older adults to evaluate the impact of the occupational therapy intervention on the primary outcomes of frailty status and physical functioning, and the secondary outcomes of occupational performance, health status, quality of life and care usage. Hypotheses: Frailty status and physical functioning will be significantly improved following the intervention and will be maintained for 6-months after treatment termination.

ELIGIBILITY:
Inclusion Criteria:

* Prefrail (meeting 1-2 of the following 5 criteria: self-report of loss of at least 10% of body weight over a 2-year period and the four following questions: (1) "Because of health problems, do you have any difficulty with lifting or carrying weights over 10 pounds, like a heavy bag of groceries?", (2) "Because of a health problem, do you have any difficulty with getting up from a chair after sitting for long periods?", (3) "Have you had any of the following persistent or troublesome problems: severe fatigue or exhaustion?", and (4) "Have you fallen down in the past 2 years?" )
* African American
* Age 55 and older

Exclusion Criteria:

* Moderate to severe dementia
* A serious physical disability that requires a caregiver to provide care for basic activities of daily living
* A terminal illness (e.g., end stage renal disease or end stage cancer).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Habit formation | from week 0 to week 4
  Self-reported Behavioral Automaticity index
Frailty | From week 0 to week 16
  Fried Frailty Index

SECONDARY OUTCOMES:
Self Rate Quality of Life | From week 0 to week 16
  WHOQOL BREF (brief version)
Social Participation | From week 0 to week 16
  NIH PROMISE Ability to Participate & Satisfaction with Social Roles (Short forms 8a)
Global Health | From week 0 to week 16
  NIH PROMISE Global Health form
Health Service Utilization | From week 0 to week 40
  Narrative self-report of services

CONTACTS AND LOCATIONS:
Overall Officials: Heather Fritz, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No